CLINICAL TRIAL: NCT06170151
Title: Role of18F-FDG PET-CT for Assessing and Predicting Response to Daratumumab and for Prognosis With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: DaRMy PET
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic accuracy — evaluate the role of 18F-FDG PET-CT for assessing early response after 6 months of treatment in patients with relapsed/refractory multiple myeloma.

SUMMARY:
Positron Emission Tomography - Computed Tomography (PET-CT) using fluorine-18 fluorodeoxyglucose is a functional imaging diagnostic tool which is widely used In several neoplastic conditions, at initial staging, for restaging in suspected disease relapse and for assessing the response to treatment. Most patients with multiple myeloma (MM) exhibit a high-glycolytic activity rate and therefore they are FOG-avid, especially at the disease relapse. The priceless value of 18F-FOG PET-CT in the therapeutic assessment for several treatment schemes, including aSCT, has been highlighted by several studies: particularly, the occurrence of negative PET-CT after a double aSCT in MM patients with clinical complete response or very good partial response positively correlates with favourable PFS and overall survival (OS). likewise, persistence of 18F-FDG avid disease in MM patients achieving a clinical complete response constitutes a poor prognostic factor. Primary objective of this prospective, observational, non-pharmacological, multicentric study is to evaluate the role of 18F-FDG PET-CT for assessing early response after 6 months of treatment with daratumumab in patients with .relapsed/refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* patients with refractory multiple myeloma who relapsed after therapy with daratumumab in combination with dexamethasone + bortezomib or dexamethasone + lenalidomide;
* patients capable of expressing informed consent.

Exclusion Criteria:

* patients with clinical contraindications to the administration of daratumumab;
* patients with coexisting non-hematological neoplastic condition;
* patients< 18 years;
* patients uncapable of expressing informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with refractory multiple myeloma who relapsed after therapy with daratumumab in combination with dexamethasone + bortezomib or dexamethasone + lenalidomide.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
18F-FDG PET-CT to predicting response to treatment and to predicting prognosis in patients with relapsed/refractory multiple myeloma. | 1 year
  Positron Emission Tomography - Computed Tomography (PET-CT) using fluorine-18 fluorodeoxyglucose to assess early response after 6 months of treatment with daratumumab in 10 patients with relapsed/refractory multiple myeloma.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No